CLINICAL TRIAL: NCT03753269
Title: Efficacy of Early Intracoronary Administration of Fasudil Hydrochloride on Myocardial Perfusion in the Primary PCI of ST-elevation Myocardial Infarction: an Prospective, Randomized and Multicenter Trial
Brief Title: Early Intracoronary Administration of Fasudil in the Primary PCI of ST-segment-Elevation Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EARLY-MYO-FASUDIL
Record Dates: First submitted 2018-11-16; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: myocardial infarction; reperfusion therapy; microvascular dysfunction; Fasudil Hydrochloride; myocardial perfusion
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — fasudil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasudil Hydrochloride (Experimental): Fasudil Hydrochoride will be delivered into culprit vessel right after the first wire passage
  Interventions: Drug: Fasudil Hydrochloride
- Placebo saline (Placebo Comparator): Same volume of 0.9% saline will be delivered into culprit vessel right after the first wire passage
  Interventions: Drug: Placebo saline

INTERVENTIONS:
Drug: Fasudil Hydrochloride — 2.5mg fasudil hydrochloride (diulted to 15ml by 0.9% saline )will be delivered by targeted perfusion micro-catheter into culprit vessel right after the first wire passage
  Arms: Fasudil Hydrochloride
Drug: Placebo saline — 15ml 0.9% saline will be delivered by targeted perfusion micro-catheter into culprit vessel right after the first wire passage
  Arms: Placebo saline

SUMMARY:
The study aims to evaluate whether an early intracoronary administration of Fasudil Hydrochloride during primary PCI of STEMI can improve epicardial and myocardial perfusion as well as clinical outcomes.

DETAILED DESCRIPTION:
Timely reperfusion therapy is the most effective treatment for acute STEMI patients. Primary PCI has been documented as the best method for restoration of epicardial blood flow. Nevertheless, recovery of epicardial blood flow does not necessarily equate to a sufficient reperfusion at myocardial level. Although epicardial TIMI 3 flow could be achieved in the majority of STEMI patients by contemporary PPCI, it has been well acknowledged that microvascular obstruction (MVO) is far more prevalent than the epicardial no-reflow phenomenon and has huge detrimental impact on clinical outcomes.

Routine thrombus aspiration by special catheter during primary PCI has shown negative or even harmful results in clinical trials. Distal coronary protective devices are also ineffective to improve myocardial perfusion. On the contrary, peri-procedual administration of several medications has shown possibilities to reduce MVO. These medications are mostly anti-platelet agents such as GP IIb/IIIa receptor and microvascular dilators like adenosine, sodium nitroprusside and verapamil. Theoretically, intracoronary delivery of medications can be more effective and potentially decrease side effects. Empirical application of aforementioned agents seems to improve the epicardial flow in patients not achieving TIMI 3 flow after PCI. However, it is debatable whether early administration of intracoronary medication (meaning before PCI) may further reduce MVO assuming it could be better to reduce reperfusion injury. However, this has not been well investigated yet.

Rho-associated protein kinase (Rho kinase) is expressed in many cells, including smooth muscle cells and vascular endothelial. Activation of Rho kinase leads to increased smooth muscle intracellular calcium and robust vasoconstriction. Fasudil hydrochloride is a rho-kinase inhibitor that severs clinically as a potent small vessel dilator, especially in the field of cerebral circulation. Meanwhile, It has been empirically used in individual STEMI cases and showed effectiveness in improving coronary flow for PCI therapy. This study aims to evaluate whether an early intracoronary administration of Fasudil Hydrochloride can improve myocardial perfusion and clinical outcomes for STEMI patients undergoing primary PCI. To ensure the complete delivery of agents within coronary, a special-designed targeted perfusion micro-catheter will be used for drug delivery. Patients in the control arm will be administrated by intracoronary saline.

For the results, coronary angiography-based index of epical and myocardial perfusion will be analyzed. MVO will be determined by cardiac magnetic resonance imaging and quantified as the percentage of left ventricular myocardial mass (% LV). The rate of composite major adverse cardiac events (MACEs) at 30 days and 6 months since symptom onset will be the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 or 18 years old, less than 75 years old;

  * Patents with myocardial infarction who have symptom onset within 6h before randomization;
  * ECG: ≥2 mm ST-segment elevation in 2 contiguous precordial leads or ≥1 mm ST-segment elevation in 2 contiguous extremity leads ;
  * Signed informed consent form prior to trial participation

Exclusion Criteria:

1. ECG with new left bundle branch block;
2. Contraindications for CMR
3. Repeated STEMI
4. History of cardiovascular diseases

   * PCI within previous 1 month or Previous coronary-artery bypass surgery (CABG)
   * Previously known multi-vessel coronary artery disease not suitable for revascularization
   * Hospitalization for cardiac reason within past 48 hours
   * Known acute pericarditis and/or subacute bacterial endocarditis
   * Arterial aneurysm, arterial/venous malformation and aorta dissection;
5. History of other severe diseases

   * Any other diseases with life expectancy ≤12 months
   * • Any history of severe renal or hepatic dysfunction (hepatic failure, cirrhosis, portal hypertension and active hepatitis); Neutropenia, thrombocytopenia; Known acute pancreatitis
6. Severe cardiac complications

   * Any sign of cardiac rupture
   * Cardiogenic shock (SBP <90 mmHg after fluid infusion or SBP<100 mmHg after vasoactive drugs)
7. Not suitable for clinical trial

   * Inclusion in another clinical trial;
   * Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 7 days;
   * Pregnancy or lactating;
   * Body weight <40kg or >125kg;
   * Known allergy to any drug that may appear in the study
   * Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete epicardial and myocardial reperfusion after PCI | PCI procedure
  The percentage of patient achieving both thrombolysis in myocardial infarction (TIMI) flow grade (TFG) 3 for epicardial reperfusion and TIMI myocardial perfusion (TMPG) grade 3 for myocardial reperfusion
CMR-derived microvascular obstruction (MVO) | Within one week after the STEMI onset
  MVO is defined as hypoenhanced area within infracted zone presented by CMR gadolinium late enhancement imaging. MVO will be quantified as the percentage of LV mass (% LV)

SECONDARY OUTCOMES:
CMR-derived infarction size | Within one week of STEMI onset, repeated on the sixth month
  Infarct size was determined by the extent of late gadolinium enhancement on CMR and expressed as a percentage of LV mass (% LV)
TIMI Flow Grade (TFG) | PCI procedure
  Percentage of patients achieving TFG 3
TIMI Myocardial Perfusion Grade (TMPG) | PCI procedure
  Percentage of patients achieving TMPG 3
TMPFC | PCI procedure
  Mean or median value of TMPFC
Complete ST-segment Resolution | 90 minutes after PCI procedure
  Percentage of patients achieving ≥ 70% resolution of the initial sum of ST-segment elevation
MACEs | 30 days and 6 months after STEMI onset
  Incidence of major adverse cardiac events (MACEs) as a composite of all cause death, nonfatal reinfarction, heart failure and stroke after PCI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding S, Pu J, Qiao ZQ, Shan P, Song W, Du Y, Shen JY, Jin SX, Sun Y, Shen L, Lim YL, He B. TIMI myocardial perfusion frame count: a new method to assess myocardial perfusion and its predictive value for short-term prognosis. Catheter Cardiovasc Interv. 2010 Apr 1;75(5):722-32. doi: 10.1002/ccd.22298. PMID 19960517
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197
- [Background] Kidambi A, Mather AN, Motwani M, Swoboda P, Uddin A, Greenwood JP, Plein S. The effect of microvascular obstruction and intramyocardial hemorrhage on contractile recovery in reperfused myocardial infarction: insights from cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 Jun 27;15(1):58. doi: 10.1186/1532-429X-15-58. PMID 23806080
- [Background] Taniguchi Y, Funayama H, Matsuda J, Fujita K, Nakagawa T, Nakamura T, Umemoto T, Mitsuhashi T, Ako J, Momomura S. Super-selective intracoronary injection of Rho-kinase inhibitor relieves refractory coronary vasospasms: a case report. Int J Cardiol. 2014 Sep;176(1):270-1. doi: 10.1016/j.ijcard.2014.06.096. Epub 2014 Jul 8. No abstract available. PMID 25065335
- [Background] TIMI Study Group. The Thrombolysis in Myocardial Infarction (TIMI) trial. Phase I findings. N Engl J Med. 1985 Apr 4;312(14):932-6. doi: 10.1056/NEJM198504043121437. No abstract available. PMID 4038784
- [Background] Masumoto A, Hirooka Y, Shimokawa H, Hironaga K, Setoguchi S, Takeshita A. Possible involvement of Rho-kinase in the pathogenesis of hypertension in humans. Hypertension. 2001 Dec 1;38(6):1307-10. doi: 10.1161/hy1201.096541. PMID 11751708
- [Background] Uehata M, Ishizaki T, Satoh H, Ono T, Kawahara T, Morishita T, Tamakawa H, Yamagami K, Inui J, Maekawa M, Narumiya S. Calcium sensitization of smooth muscle mediated by a Rho-associated protein kinase in hypertension. Nature. 1997 Oct 30;389(6654):990-4. doi: 10.1038/40187. PMID 9353125